CLINICAL TRIAL: NCT03323736
Title: A Prospective, Single-arm, Multicenter Study to Evaluate Effectiveness and Safety of Tympanostomy Tube Placement Using the Tula Iontophoresis and Tube Delivery Systems for Children in an Office Setting.
Brief Title: In-Office Tympanostomy Tube Placement in Children (OTTER)
Acronym: OTTER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tusker Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR007001
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Results first posted 2020-01-31 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: OME - Otitis Media With Effusion; AOM - Acute Otitis Media
MeSH Terms: conditions — Otitis Media with Effusion; Otitis Media | interventions — Iontophoresis

STUDY DESIGN:
Intervention Model Description: Pivotal cohort is single arm. Physician initial subjects evaluated in separate cohorts but not included in primary and secondary analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Pivotal Cohort (Other): Active Tymbion iontophoresis and tube insertion using the Tube Delivery System in-office.
  Interventions: Combination Product: Iontophoresis & tube placement
- Office Lead-In Cohort (Other): Active Tymbion iontophoresis and tube insertion using the Tube Delivery System in-office. Physician initial in-office iontophoresis and tube insertion procedures (minimum of 2 subjects per investigator).
  Interventions: Combination Product: Iontophoresis & tube placement
- OR Lead-In Cohort (Other): Tubes insertion using the Tube Delivery System in the operating room (OR). Physician initial tube insertion procedures in the OR (minimum of 2 subjects per investigator).
  Interventions: Device: Tube placement

INTERVENTIONS:
Combination Product: Iontophoresis & tube placement — Subjects will receive active Tymbion iontophoresis and will have tubes placed in-office using the Tube Delivery System in all ears indicated for tube placement.
  Arms: Office Lead-In Cohort; Pivotal Cohort
Device: Tube placement — Subjects will have tubes placed in the OR using the Tube Delivery System in all ears indicated for tube placement.
  Arms: OR Lead-In Cohort

SUMMARY:
A prospective, single-arm, multicenter study to evaluate effectiveness and safety of Tymbion iontophoresis and tympanostomy tube placement using the Tula Iontophoresis and Tube Delivery Systems for children in an office setting.

DETAILED DESCRIPTION:
The objective of this study is to evaluate effectiveness and safety of tympanostomy tube (TT) placement in children following local anesthesia in a physician's clinic setting (henceforth referred to as 'in-office'). Local anesthesia using Tymbion, a lidocaine-based anesthetic, is delivered by the Tula Iontophoresis System (IPS) and TT placement is implemented by the Tula Tube Delivery System (TDS).

The IPS will be used to facilitate anesthetic delivery to the tympanic membrane (TM). The Iontophoresis System consists of an Iontophoresis Control Unit, Iontophoresis Earsets and a return electrode patch. The Control Unit monitors and delivers a fixed amount of charge (ie, dose) to the patient through the Earsets(s) and alerts the operator when charge delivery is complete. The lidocaine-based solution used for local anesthesia of the TM is Tymbion (2% lidocaine HCl/ 1:100,000 epinephrine).

The TDS is a mechanical device that integrates a myringotomy blade, tympanostomy tube and tube inserter for TT placement with a user-controlled activation. The study will use the TDS with a grommet-type tube.

This pivotal study will include up to 422 children ages 6 months through 12 years indicated for tympanostomy tube placement enrolled at approximately 15 to 25 investigational centers in the US and Canada. The pivotal cohort consists of 222 subjects. In addition, up to 100 subjects will be enrolled as lead-in procedures in the OR using the TDS and up to 100 subjects will be enrolled as lead-in procedure in-office (using IPS and TDS) as the surgeons' initial experience with the technology prior to enrolling into the pivotal cohort.

All pivotal and lead-in subjects will follow the same study protocol assessments and visit schedule consisting of a screening visit, procedure visit and 3-week, 6 month, 12 month, 18 month, and 24 month post-procedure follow-up visits. Lead-in procedures will be analyzed separately from the pivotal pediatric cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females at least 6 months old through 12 years old at time of consent
2. Indication for tympanostomy tube insertion per Clinical Practice Guideline
3. Behavioral capacity and cooperative temperament to undergo an awake procedure, based on physician judgment (not applicable to OR Lead-In subjects)
4. Subject's parent/guardian and subject are able and willing to comply with the protocol and attend all study visits
5. Subject's parent/guardian and subject are able and willing to provide informed consent or assent as age appropriate

Exclusion Criteria:

1. Significantly atrophic, retracted, bimeric, monomeric or atelectatic tympanic membrane
2. Perforated tympanic membrane
3. Otitis externa
4. Active or recent conditions of the tympanic membrane (eg, prior myringotomy with incomplete wound healing or re-epithelization)
5. Hemotympanum
6. Damaged/denuded skin in the auditory canal
7. Cerumen impaction resulting in a significant amount of cleaning required to visualize the tympanic membrane potentially causing abrasion or irritation to the external ear canal
8. Anatomy that precludes sufficient visualization of and access to the tympanic membrane
9. Anatomy that necessitates tympanostomy tube placement in the posterior half of the tympanic membrane
10. History of sensitivity or allergic reaction to lidocaine HCl, tetracaine, epinephrine, or any hypersensitivity to local anesthetics of the amide type, or any component of the anesthetic drug formulation (not applicable to OR Lead-In subjects)
11. Familial history of insensitivity to lidocaine or other local anesthetics of the amide type (eg, history of inadequate anesthesia with dental numbing agents). (not applicable to OR Lead-In subjects)
12. Electrically sensitive medical support systems (eg, pacemakers, defibrillators, cochlear implants)
13. Other conditions that would preclude performing the study procedure including iontophoresis system ear plug incompatibility.
14. Health conditions that, in the opinion of the investigator, would present undue risk to the subject, based on device/anesthetic drug product label warnings and precautions.
15. Subject is 4 years or older and not able to complete all baseline assessments. Subject is younger than 4 years and not able to complete all baseline assessments, not including audiometry.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 370 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2021-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lustig, Principal Investigator — Columbia University
Locations (19):
- United States (18):
  - California Head and Neck Specialists, Carlsbad, California
  - Sacramento ENT, Roseville, California
  - Camino Ear Nose & Throat Clinic, San Jose, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale School of Medicine, Section of Otolaryngology, New Haven, Connecticut
  - South Florida Pediatric Otolaryngology, Fort Lauderdale, Florida
  - Nemour's Children's Specialty Care, Jacksonville, Florida
  - Advanced ENT & Allergy, Louisville, Kentucky
  - Albany ENT & Allergy Services, Albany, New York
  - Columbia University Medical Center, New York, New York
  - Charlotte Ear Eye Nose & Throat Associates, PA, Charlotte, North Carolina
  - Specialty Physician Associates, Bethlehem, Pennsylvania
  - South Carolina Ear Nose and Throat, Lugoff, South Carolina
  - Carolina Ear Nose and Throat Clinic, Orangeburg, South Carolina
  - Ear Nose and Throat Specialists of Abilene, Abilene, Texas
  - Frisco ENT for Children, Frisco, Texas
  - Collin County ENT, Frisco, Texas
  - Ear Medical Group, San Antonio, Texas
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pivotal Cohort: Active Tymbion iontophoresis and tube insertion in all ears indicated for tube placement using the Tube Delivery System (TDS) in office.
- Office Lead-In Cohort: Active Tymbion iontophoresis and tube insertion in all indicated ears using the Tube Delivery System in-office. Physician initial iontophoresis and tube insertion procedures (minimum of 2 subjects per investigator).
- OR Lead-In Cohort: Tube insertion using the Tube Delivery System (TDS) in all indicated ears in the operating room (OR). Physician initial tube insertion procedures using the TDS in the OR (minimum of 2 subjects per investigator).
Period: Overall Study
Arm/Group | Pivotal Cohort | Office Lead-In Cohort | OR Lead-In Cohort
Started | 241 | 59 | 70
Treated | 222 | 47 | 68
Completed | 222 | 47 | 68
Not Completed | 19 | 12 | 2
Not completed — Screen Failure | 14 | 9 | 1
Not completed — Withdrawal Before Treatment | 3 | 1 | 1
Not completed — Iontophoresis fill/no iontophoresis | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pivotal Cohort | Office Lead-In Cohort | OR Lead-In Cohort | Total
Number analyzed (Participants) | 222 | 47 | 68 | 337
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.7 (3.18) | 4.8 (3.10) | 3.4 (2.55) | 4.5 (3.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 20 | 28 | 141
  Male | 129 | 27 | 40 | 196
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 6 | 14 | 51
  Not Hispanic or Latino | 191 | 40 | 54 | 285
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 0 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 24 | 6 | 6 | 36
  White | 183 | 35 | 53 | 271
  More than one race | 4 | 1 | 0 | 5
  Unknown or Not Reported | 7 | 5 | 6 | 18
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 4 | 4 | 11
  United States | 219 | 43 | 64 | 326

OUTCOME MEASURES:

1. Primary Outcome: Procedural Success:
Description: Count (and percentage) of subjects in the pivotal cohort with successful placement of Tusker Medical tympanostomy tubes in all indicated ears in an office procedure. Note: the primary endpoint applies only to the Pivotal Cohort, and not to the OR Lead-In or Office Lead-In cohorts.
Time Frame: Day of Procedure (Day 0) Immediately following tube placement
Measure: Count of Participants; unit: Participants
Groups:
- Pivotal Cohort (6 Month to <5 Year Old Children); Pivotal Cohort (5 Through 12 Year Old Children): Active Tymbion iontophoresis and tubes insertion using the Tube Delivery System in-office
  Iontophoresis & tube placement: Subjects will receive active Tymbion iontophoresis and will have tubes placed in-office using the tube delivery system in all ears indicated for tube placement.
Arm/Group | Pivotal Cohort (6 Month to <5 Year Old Children) | Pivotal Cohort (5 Through 12 Year Old Children)
Number analyzed (Participants) | 120 | 102
Participants | 103 | 91
Statistical Analysis 1: Comparison: Pivotal Cohort (6 Month to <5 Year Old Children); Procedural success rate was compared to the performance goal of 68% using a Bayesian Hierarchical model; Test type: Superiority — The Procedural Success endpoint would be successfully met if the lower bound of the 95% Credible Interval (lower limit 0.80) exceeded the 68% success rate performance goal; Credible Interval = 0.86, 95% CI 2-sided [0.80 to 0.91]
Statistical Analysis 2: Comparison: Pivotal Cohort (5 Through 12 Year Old Children); Procedural success rate was compared to the performance goal of 68% using a Bayesian Hierarchical model; Test type: Superiority — The Procedural Success endpoint would be successfully met if the lower bound of the 95% Credible Interval (lower limit 0.82) exceeded the 68% success rate performance goal; Credible Interval = 0.89, 95% CI 2-sided [0.82 to 0.93]

2. Primary Outcome: Tube Placement Tolerability
Description: Mean subject-reported pain score following TDS tube placement using the Faces Pain Scale-Revised (FPS-R) (pivotal cohort children ages 5 and older only). The FPS-R has 6 faces which permits scaling to a 0-to-10 scoring system in intervals of 2 (ie 0, 2, 4, 6, 8 and 10), where 0 represents 'no pain' and 10 represents 'very much pain'. Note- the primary endpoint applies only to the Pivotal Cohort, and not to the OR Lead-In or Office Lead-In cohorts.
Time Frame: Day of Procedure (Day 0) Immediately following tube placement
Population: Subjects with successful tube placement only. Note - 2 subjects were excluded from analysis because they did not self-report their pain scores, resulting in 89 participants analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pivotal Cohort (5 Through 12 Year Olds): Active Tymbion iontophoresis and tubes insertion using the Tube Delivery System in-office
  Iontophoresis & tube placement: Subjects will receive active Tymbion iontophoresis and will have tubes placed in-office using the tube delivery system in all ears indicated for tube placement.
Arm/Group | Pivotal Cohort (5 Through 12 Year Olds)
Number analyzed (Participants) | 89
score on a scale | 3.30 (3.39)
Statistical Analysis 1: Comparison: Pivotal Cohort (5 Through 12 Year Olds); Test type: Superiority — Comparison of mean tube placement FPS-R score to a performance goal of 4.2; p = 0.0072, t-test, 1 sided — Mean FPS-R score hypothesized to be less than (superior to) a performance goal of 4.2, at a significance level of 0.025 (p<0.025)

3. Secondary Outcome: Tube Patency
Description: Count (and percentage) of subjects in the pivotal cohort, in which a Tusker Medical tube was successfully placed, with functionally patent tube(s) at the 3-week post-procedure follow-up visit.
  Note- thus secondary endpoint applies only to the Pivotal Cohort, and not to the OR Lead-In or Office Lead-In cohorts.
  Note - This endpoint includes subjects for which at least 1 ear had successful tube placement. For bilateral subjects, they may be considered a non-successful procedure if only 1 ear had successful tube placement, however would be evaluated for the Tube Patency endpoint for the ear that was successful.
Time Frame: 3 Weeks Post Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Pivotal Cohort
Number analyzed (Participants) | 208
Participants | 191
Statistical Analysis 1: Comparison: Pivotal Cohort; Tube Patency endpoint would be successfully met if the percentage of subjects with patent tubes was greater than (superior to) 80% (by subject), at a significance level of 0.025 (p<0.025); Test type: Superiority; p < 0.0001, mid-P method for single proportion — Pre-specified threshold for superiority was >80%, at alpha = 0.025

4. Secondary Outcome: Tube Retention
Description: Count (percentage) of subjects in the pivotal cohort, in which a Tusker Medical tube(s) was successfully placed, with presence of a Tusker Medical tube across the TM in all successfully treated ears at the 3-week post-procedure follow-up visit.
  Note- the secondary endpoint applies only to the Pivotal Cohort, and not to the OR Lead-In or Office Lead-In cohorts.
  Note - This endpoint includes subjects for which at least 1 ear had successful tube placement. For bilateral subjects, they may be considered a non-successful procedure if only 1 ear had successful tube placement, however would be evaluated for the Tube Retention endpoint for the ear that was successful.
Time Frame: 3 Weeks Post Procedure
Measure: Count of Participants; unit: Participants
Groups:
- Pivotal Cohort: Active Tymbion iontophoresis and tubes insertion using the Tube Delivery System in-office
  Iontophoresis & tube placement: Subjects will receive active Tymbion iontophoresis and will have tubes placed in-office using the tube delivery system in all ears indicated for tube placement.
Arm/Group | Pivotal Cohort
Number analyzed (Participants) | 208
Participants | 206
Statistical Analysis 1: Comparison: Pivotal Cohort; Tube Retention endpoint would be successfully met if the percentage of subjects with retained tubes was greater than (superior to) 88% (by subject), at a significance level of 0.025 (p<0.025); Test type: Superiority; p < 0.0001, mid-P method for single proportion — Pre-specified threshold for superiority was >88%, at alpha = 0.025

5. Secondary Outcome: Anesthesia Effectiveness
Description: Count (percentage) of subjects in the pivotal cohort, who completed iontophoresis for all indicated ears, with adequate anesthesia for TT placement in all treated ears as determined by physician's evaluation of TM anesthesia prior to tube placement.
  Note- the secondary endpoint applies only to the Pivotal Cohort, and not to the OR Lead-In or Office Lead-In cohorts.
Time Frame: Day of Procedure (Day 0)
Measure: Count of Participants; unit: Participants
Arm/Group | Pivotal Cohort
Number analyzed (Participants) | 220
Participants | 206
Statistical Analysis 1: Comparison: Pivotal Cohort; The Anesthesia Effectiveness endpoint would be successfully met if the percentage of subjects with successful anesthesia was greater than (superior to) 85% (by subject), at a significance level of 0.025 (p<0.025); Test type: Superiority; p < 0.0001, mid-P method for single proportion — Pre-specified threshold for superiority was >85%, at alpha = 0.025

ADVERSE EVENTS:
Time Frame: Procedure through most recent follow-up visit with mean follow-up of 14.3 months (all cohorts combined). Individual cohort mean follow-up time is 11.3 months for OR Lead-In Cohort, 14.1 months for Office Lead-In Cohort, and 15.3 months for Pivotal Cohort.
Groups:
- OR Lead-In Cohort (Subjects Treated in OR): Tube insertion using the Tube Delivery System (TDS) in all indicated ears in the operating room (OR). Physician initial tube insertion procedures using the TDS in the OR (minimum of 2 subjects per investigator).
- Office Lead-In Cohort (Subjects Treated in Office): Active Tymbion iontophoresis and tube insertion in all ears indicated for tube placement using the Tube Delivery System (TDS) in office. Physician initial tube insertion procedures using the Iontophoresis System and the TDS in the Office (minimum of 2 subjects per investigator).
- Pivotal Cohort (Subjects Treated in Office): Active Tymbion iontophoresis and tube insertion in all ears indicated for tube placement using the Tube Delivery System (TDS) in office.
Arm/Group | OR Lead-In Cohort (Subjects Treated in OR) | Office Lead-In Cohort (Subjects Treated in Office) | Pivotal Cohort (Subjects Treated in Office)
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/47 | 0/222
Serious Adverse Events (participants affected / at risk) | 4/68 | 0/47 | 3/222
Other Adverse Events (participants affected / at risk) | 28/68 | 22/47 | 79/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OR Lead-In Cohort (Subjects Treated in OR) (N=68) | Office Lead-In Cohort (Subjects Treated in Office) (N=47) | Pivotal Cohort (Subjects Treated in Office) (N=222)
Respiratory Syncytial Virus Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) — Not related to device, drug or procedure
Wrist Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device, drug or procedure
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to device, drug or procedure
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to device, drug or procedure
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) — Not related to device, drug or procedure
Velopharyngeal Insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device, drug or procedure
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OR Lead-In Cohort (Subjects Treated in OR) (N=68) | Office Lead-In Cohort (Subjects Treated in Office) (N=47) | Pivotal Cohort (Subjects Treated in Office) (N=222)
Inadequate Anesthesia (Ear and labyrinth disorders) | 0 (0) | 4 (4) | 8 (8) — Inadequate anesthesia determined after completion of Tymbion iontophoresis procedure and prior to attempting tube placement. Potentially related to device, drug or procedure. This event type is not applicable to OR procedures.
Occluded Tube (Ear and labyrinth disorders) | 13 (15) | 5 (6) | 51 (65) — 2 events for 2 OR subjects and 6 events for 6 Pivotal subjects considered potentially related to device or procedure. All other Occluded Tube events considered not related to device, drug or procedure.
Otorrhea (Ear and labyrinth disorders) | 19 (29) | 7 (14) | 60 (97) — 1 event for 1 OR subject considered potentially related to procedure. All other Otorrhea events not related to device, drug or procedure.
Ear Pain (Ear and labyrinth disorders) | 6 (6) | 9 (9) | 29 (32) — 1 event for 1 Office Lead-In subject and 1 event for 1 Pivotal subject considered related to procedure. All other Ear Pain events considered not related to device, drug or procedure.
Otitis Media (Ear and labyrinth disorders) | 13 (25) | 11 (14) | 61 (77) — Not related to device, drug or procedure
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 3 (3) | 18 (21) — Not related to device, drug or procedure
Acute Sinusitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (2) | 16 (18) — Not related to device, drug or procedure
Pharyngitis Streptococcal (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 17 (17) — Not related to device, drug or procedure
Ear infection (Ear and labyrinth disorders) | 6 (9) | 4 (7) | 12 (15) — Not related to device, drug or procedure
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 4 (13) | 10 (14) — Not related to device, drug or procedure
Croup (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0) | 2 (3) — Not related to device, drug or procedure
Middle ear effusion (Ear and labyrinth disorders) | 2 (2) | 4 (6) | 15 (15) — Not related to device, drug or procedure
Otitis externa (Ear and labyrinth disorders) | 1 (1) | 3 (10) | 7 (8) — Not related to device, drug or procedure
Fever (General disorders) | 0 (0) | 3 (3) | 6 (7) — Not related to device, drug or procedure
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 6 (6) — Not related to device, drug or procedure
Influenza (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 6 (6) — Not related to device, drug or procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must submit communications to Sponsor for review and comment to verify accurate content at least 30 days prior to submitting to any third party. A delay up to 90 days may be requested by Sponsor in order to file patent applications relating to an Invention if applicable. Sponsor and PI agree that any Institution Publication shall only be made after the Multicenter Publication, provided that the Multicenter Publication is submitted within 18 months after conclusion of the study at all sites.

DOCUMENTS (2):
  • Study Protocol (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT03323736/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT03323736/SAP_001.pdf